CLINICAL TRIAL: NCT04817800
Title: An Open Label, Randomized, Three-treatment, Three-period, Crossover, Single Dose Study, to Investigate Drug-drug Interaction and Relative Bioavailability Between the Fixed Dose Combination Azelastine Hydrochloride / Beclomethasone Dipropionate (140/100 μg Azelastine Hydrochloride / Beclomethasone Dipropionate) Nasal Spray, and Beclomethasone Dipropionate Nasal Spray (100 μg Beclomethasone Dipropionate) in the Test Vehicle, and the Commercially Available Product, RinoClenil® Nasal Spray (100 μg Beclomethasone Dipropionate), in Healthy Subjects Under Fasting Conditions
Brief Title: To Investigate Drug-drug Interaction and Relative Bioavailability Between the FDC AzelastineHCL/Beclomethasone Dipropionate Nasal Spray, & Beclomethasone Dipropionate Nasal Spray in the Test Vehicle, and RinoClenil® Nasal Spray
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 980-2020
Record Dates: First submitted 2021-03-19; First posted 2021-03-26 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine; Beclomethasone; Nasal Sprays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 140/100 μg Azelastine hydrochloride/Beclomethasone Dipropionate) (Experimental)
  Interventions: Drug: 140/100 μg Azelastine hydrochloride/Beclomethasone Dipropionate)
- 100 μg Beclomethasone dipropionate, Nasal Spray (Experimental)
  Interventions: Drug: 140/100 μg Azelastine hydrochloride/Beclomethasone Dipropionate)
- RinoClenil® Nasal Spray (100 μg Beclomethasone Dipropionate) (Active Comparator)
  Interventions: Drug: 140/100 μg Azelastine hydrochloride/Beclomethasone Dipropionate)

INTERVENTIONS:
Drug: 140/100 μg Azelastine hydrochloride/Beclomethasone Dipropionate) — It will be nasaly administered
  Other Names: 100 μg Beclomethasone dipropionate, Nasal Spray; RinoClenil® Nasal Spray (100 μg Beclomethasone Dipropionate)

SUMMARY:
An open label, randomized, three-treatment, three-period, crossover, single dose study, to investigate drug-drug interaction and relative bioavailability between the fixed dose combination Azelastine hydrochloride / Beclomethasone dipropionate (140/100 μg Azelastine hydrochloride / Beclomethasone dipropionate) Nasal Spray, and Beclomethasone Dipropionate Nasal Spray (100 μg Beclomethasone Dipropionate) in the test vehicle, and the commercially available product, RinoClenil® Nasal Spray (100 μg Beclomethasone Dipropionate), in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* The subject is Caucasian & aged between eighteen & fifty years (18 - 50), both inclusive.
* The subject is within the limits for his height & weight as defined by the body mass index range
* (18.5 - 30.0 Kg/m2).
* The subject is willing to undergo the necessary pre- & post- medical examinations set by this
* study.
* The results of medical history, vital signs, physical examination & conducted medical laboratory
* tests are normal as determined by the clinical investigator.
* The subject tested negative for hepatitis (HBsAg, HCVAb) viruses and human immunodeficiency
* virus (HIVAb).
* There is no evidence of psychiatric disorder, antagonistic personality and poor motivation,
* emotional or intellectual problems likely to limit the validity of consent to participate in the study
* or limit the ability to comply with protocol requirements.
* The subject is able to understand and willing to sign the informed consent form.
* For female subjects: negative pregnancy test and the woman is using two reliable contraception
* methods & should be non-lactating.
* The subject has normal cardiovascular system and ECG recording.
* The subject kidney and liver (AST & ALT enzymes) functions tests are within normal range.

Exclusion Criteria:

* The subject is smoker/ has positive cotinine test.
* The subject has suffered an acute illness one week before dosing.
* The subject has a history of or concurrent abuse of alcohol.
* The subject has a history of or concurrent abuse of illicit drugs.
* The subject has a history of hypersensitivity and/or contraindications to the study drug, its
* excipients and any related compounds.
* The subject has been hospitalized within three months before the study or during the study.
* The subject is vegetarian.
* The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days
* before dosing and until 23 hours after dosing in all study periods.
* The subject has taken a prescription medication within two weeks or even an over the counter
* product (OTC) within one week before dosing in each study period and any time during the study,
* unless otherwise judged acceptable by the clinical investigator.
* The subject has taken grapefruit containing beverages or foodstuffs within seven (7) days before
* first dosing and any time during the study.
* The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and
* bioequivalence studies) within the last 80 days prior to the present study.
* The subject has donated blood within 80 days before first dosing.
* The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal,
* hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or
* psychiatric diseases.
* The subject has consumed drugs that may affect pharmacological or pharmacokinetic properties
* (ritonavir, cobicistat & CNS depressants) two weeks before dosing, during the study and two
* weeks after dosing.
* The subject has recent nose surgery or a history of chronic sinusitis, recent URTI and nasal septum
* deviation that may affect nasal mucosa integrity.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of Beclomethasone dipropionate and its active metabolite Beclomethasone 17-monopropionate | 23 hours
  For the assessment of a potential drug-drug interaction, no effect of Azelastine on the pharmacokinetics of Beclomethasone dipropionate and its active metabolite Beclomethasone 17-monopropionate will be concluded if the fixed dose combination Test-to-mono test GMR and the corresponding 90% CI of the ln-transformed primary pharmacokinetic parameters are within the 80.00% to 125.00% acceptance interval.
  For the assessment of the relative bioavailability, bioequivalence between Beclomethasone dipropionate drug products will be concluded if the fixed dose combination test-to-mono reference GMR and the corresponding 90% CI of the Lntransformed primary pharmacokinetic parameters are within the 80.00% to 125.00% acceptance interval.
area under the plasma concentration versus time curve (AUC) from pre-dose (time zero) to the last sampling time with quantifiable concentrations (AUC0-t) of Beclomethasone dipropionate and its active metabolite Beclomethasone 17-monopropionate | 23 hours
  For the assessment of a potential drug-drug interaction, no effect of Azelastine on the pharmacokinetics of Beclomethasone dipropionate and its active metabolite Beclomethasone 17-monopropionate will be concluded if the fixed dose combination Test-to-mono test GMR and the corresponding 90% CI of the ln-transformed primary pharmacokinetic parameters are within the 80.00% to 125.00% acceptance interval.
  For the assessment of the relative bioavailability, bioequivalence between Beclomethasone dipropionate drug products will be concluded if the fixed dose combination test-to-mono reference GMR and the corresponding 90% CI of the Lntransformed primary pharmacokinetic parameters are within the 80.00% to 125.00% acceptance interval.
AUC from time zero to infinity (AUC0-∞) of Beclomethasone dipropionate and its active metabolite Beclomethasone 17-monopropionate | 23 hours
  For the assessment of a potential drug-drug interaction, no effect of Azelastine on the pharmacokinetics of Beclomethasone dipropionate and its active metabolite Beclomethasone 17-monopropionate will be concluded if the fixed dose combination Test-to-mono test GMR and the corresponding 90% CI of the ln-transformed primary pharmacokinetic parameters are within the 80.00% to 125.00% acceptance interval.
  For the assessment of the relative bioavailability, bioequivalence between Beclomethasone dipropionate drug products will be concluded if the fixed dose combination test-to-mono reference GMR and the corresponding 90% CI of the Lntransformed primary pharmacokinetic parameters are within the 80.00% to 125.00% acceptance interval.

SECONDARY OUTCOMES:
Obtaining the Tmax (Time to reach maximum concentration) | 23 hours
  The descriptive statistics including Maximum, Minimum and Median values will be measured for Tmax.
Blood pressure (safety and tolerability) | At 1 hour pre-dosing and 2, 4, 6, 8, 12, and 23 hours post dosing,
  Clinically significant abnormal deviations. Normal range of blood pressure > 90/60 and <140/90 mmHg. Treatment will be offered to those subjects whom blood pressure drops to 90/60 mm Hg or less and the subject will be excluded in case of not responding to treatment.
Pulse (safety and tolerability) | At 1 hour pre-dosing and 2, 4, 6, 8, 12, and 23 hours post dosing,
  Clinically significant abnormal deviations. Normal range of Pulse 60-100 Bpm.
Temperature (safety and tolerability) | At 1 hour pre-dosing and 2, 6, 10, 14, 18, 22 and 23 hours post dosing,
  Clinically significant abnormal deviations. The temperature will be measured axillary, orally or using infrared thermometer, standardized across all subjects. Normal range of temperature 36.5-37.5 ºC.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gürpınar, Study Director — Humanis Saglık
Locations (1):
- ACDIMA Biocenter, Amman, Jordan